CLINICAL TRIAL: NCT06624124
Title: SimuVersity Medical Center: Pain and Opioid Management Training in Diverse Patient Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00137370; 1R41DA059281-01A1 (NIH)
Record Dates: First submitted 2024-09-25; First posted 2024-10-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: None Volunteer
Keywords: educational methods; educational software

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training using AI-powered SimuVersity Training Platform (Experimental): Students and faculty will receive training on diversity considerations in pain and opioid management via an online gamified platform with AI-powered virtual patients to apply knowledge.
  Interventions: Behavioral: Gamified Training in Diversity Considerations in the Management of Pain and Opioid Use
- Training using traditional text-base methods (Active Comparator): Students and faculty will receive training on diversity considerations in pain and opioid management via written materials and text-base case studies to apply knowledge.
  Interventions: Behavioral: Traditional Training in Diversity Considerations in the Management of Pain and Opioid Use

INTERVENTIONS:
Behavioral: Gamified Training in Diversity Considerations in the Management of Pain and Opioid Use — Use of a video game-based training platform
  Arms: Training using AI-powered SimuVersity Training Platform
Behavioral: Traditional Training in Diversity Considerations in the Management of Pain and Opioid Use — Use of a traditional text-based training platform
  Arms: Training using traditional text-base methods

SUMMARY:
This study aims to compare the effectiveness of the new educational activity/game (a novel, engaging digital-training plus interaction with virtual patients to practice skills) in meeting clinical learning objectives and outcomes compared to traditional didactic (powerpoint slide-based training and text-base case scenarios) approaches to provider and student education and satisfaction.

DETAILED DESCRIPTION:
Management of chronic pain and opioid use/misuse is challenging for clinicians and students, especially when working with diverse and underserved patient populations, and very few low-cost, flexible, highly-engaging, and effective learning resources are available to help the healthcare workforce best learn to manage these unique health concerns. Gamification holds promise as a user-friendly, fun, engaging and effective teaching strategy, especially for healthcare applications. SimuVersity Medical Center is an immersive 3D gaming platform that will engage students and practicing clinicians in a unique and captivating learning experience focused on pain and opioid management in diverse patient groups.

SimuVersity Medical Center is an innovative platform solution to education and training in specialty topics in healthcare. This novel learning platform will permit learners to explore a 3D virtual hospital space and can interact with objects, virtual colleagues/trainers and virtual patients (imbued with artificial intelligence) to learn and practice new clinical skills. The platform is built for ease-of-use with simple character controls that non-game-savvy learners find intuitive and easy. The graphical interface is clean and clear and the software runs on all modern computing platforms. The control intervention consists of traditional powerpoint slide-based training and text-base case studies for review.

This study aims to compare the effectiveness of the new educational activity/game (a novel, engaging digital-training plus interaction with virtual patients to practice skills) in meeting clinical learning objectives and outcomes compared to traditional didactic (powerpoint slide-based training and text-base case scenarios) approaches to provider and student education and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-80 years
2. English-speaking
3. Graduate-level health professional students and faculty at the Medical University of South Carolina
4. Willingness to volunteer to play the new educational game and complete questionnaires regarding satisfaction, knowledge acquisition, value, ease of use and ability to meet learning objectives

Exclusion Criteria:

1. Age outside the predefined range
2. Not a student or faculty at MUSC
3. Not willing or able to participate in the learning activity or complete study related questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Pre-Post Training Knowledge Test | From enrollment to the end of the training and assessment (2 hours later)
  Multiple-choice knowledge test on diversity considerations in pain and opioid management

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary Outcomes
Supporting Information: ICF
Time Frame: 8/31/2025
Access Criteria: Students and Faculty at the Medical University of South Carolina
URL: https://palmettoinnovations.com

DOCUMENTS (1):
  • Informed Consent Form (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT06624124/ICF_000.pdf